CLINICAL TRIAL: NCT00234299
Title: In Vivo Molecular Effects of Aspirin on Prostate Tissue
Brief Title: Effects of ASA on Prostate Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Daniel Lin, Chief of Uro-Oncology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01426-V; 05-7956-V 01 (Other: University of Washington HSD); 28526-V (Other: University of Washington HSD)
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Prostate Cancer
Keywords: Cancer; Prostate; Preventive Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Enteric coated aspirin 325mg, one tablet orally every day for six months prior to prostate biopsy.
  Interventions: Drug: Aspirin
- Group B (Placebo Comparator): Enteric coated placebo, one tablet orally every day for six months prior to prostate biopsy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — 325mg, one tablet orally, six months
  Arms: Group A
Drug: Placebo — 325mg, one tablet orally every day, 6 months
  Arms: Group B

SUMMARY:
Aspirin affects many physiological processes through its anti-inflammatory actions. Various cancers, including prostate cancer, appear to utilize inflammatory signals to facilitate their growth and progression.

We hypothesize that oral aspirin acts directly on prostate epithelial cells to alter COX-2-related metabolism and inhibit prostate cell growth.

DETAILED DESCRIPTION:
Prostate cancer is the most common non-cutaneous malignancy in men and is the second leading cause of cancer death among U.S. men. 221,000 new cases and 29,000 deaths are expected in 2003. The incidence of prostate cancer diagnosis is increasing at 3% per year. Prostate specific antigen (PSA) screening has resulted in improvements in early diagnosis of prostate cancer. However, available treatments all may have a significant negative effect on quality of life.

Studies have implicated a beneficial association between ASA use and a lower risk of other types of malignancies, including stomach, esophageal, breast, ovarian, and prostate cancer. There is significant evidence to suggest that aspirin has a protective effect against prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* May be on watchful waiting for low grade prostate cancer who are scheduled for biopsy to monitor disease.
* Have a previous diagnosis of prostatic intraepithelial neoplasia (PIN)or atypical small acinar proliferation (ASAP) before either second biopsy or even is second biopsy still has PIN or ASAP and they are to undergo a third biopsy.
* Extended-sector (at least 10 cores) prostate biopsy performed within three months of enrollment.
* Prostate tissue frozen at time of prostate biopsy (UW #04-3963-V 01)
* PSA less than 15.
* Performance status 0 or 1 by the ECOG scale.
* Ability to understand and willingness to sign an informed consent document.
* Willingness to take 325mg enteric coated aspirin daily and abstain from any other NSAID, aspirin product, or COX-2 inhibitor during the study.
* Willingness to abstain from any hormonal or herbal preparation indicated to affect hormone levels during the study.

Exclusion Criteria:

* Any prior or concurrent hormonal therapy, chemotherapy, or investigational agents.
* Use of Finasteride, Dutasteride, saw palmetto, or any herbal/nutritional preparation indicated to affect hormone levels.
* Use of 325mg aspirin three or more times a week.
* Use of NSAIDS three or more times a week.
* Use of NSAIDs, Cox-2 inhibitors and/or aspirin for 6 weeks prior to study enrollment and during the 3-month intervention.
* Known bleeding disorder.
* History of gastrointestinal bleeding.
* History of peptic or duodenal ulcer disease.
* History of stroke.
* History of serious bleeding, including but not limited to hemorrhagic stroke, epistaxis, hematuria, hematochezia, hemorrhoidal bleeding requiring cauterization.
* Uncontrolled hypertension.
* Aspirin sensitivity or allergy.
* Liver disease with known ascites, varices, clotting disorder, or liver function test >1.5 normal.
* Anemia, thrombocytopenia, prolonged INR.
* Elective surgery scheduled during 3-month intervention.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, CHD presently requiring a revascularization procedure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 45 Years to 74 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Assess the effect of oral aspirin on in vivo prostate epithelial cells. | 6 months

SECONDARY OUTCOMES:
Changes in COX-2 and COX-2 related gene expression in prostate biopsy tissue before and after the intervention; effects of the intervention on measures of apoptosis and cell cycle; effects of the intervention on global prostate gene expression. | 6 months
To measure changes in COX-2 and COX-2 related gene expression in prostate biopsy tissue before and after a 6 month intervention with enteric coated aspirin (325mg/day). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Lin, MD, Principal Investigator — Veteran's Administration Puget Sound Health Care Service
Locations (1):
- VA Puget Sound Health Care Service, Seattle, Washington, United States